CLINICAL TRIAL: NCT04192734
Title: A Retrospective Study for Evaluation of Real-world Efficacy and Safety of Ramucirumab Plus Paclitaxel in Patients With Locally-advanced Unresectable or Metastatic Gastric or Gastroesophageal Junction Adenocarcinoma
Brief Title: Retrospective Study of Ramucirumab and Paclitaxel in Gastric or Gastroesophageal Junction Adenocarcinoma
Status: Completed | Type: Observational
Sponsor: Hallym University Medical Center (Other)
Responsible Party: Principal Investigator, Zang, Dae Young, Dae Young Zang MD, PhD, Hallym University Medical Center
Other Study IDs: KCSG ST19-16
Record Dates: First submitted 2019-12-05; First posted 2019-12-10 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Gastric or Gastroesophageal Junction Adenocarcinoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a retrospective, multicenter, non-interventional study for the evaluation of real-world efficacy and safety of ramucirumab plus paclitaxel in gastric or gastroesophageal junction adenocarcinoma as part of the establishment of hospital medical record collection system to evaluate drug effectiveness by Health Insurance Review & Assessment Service (HIRA). The medical records in approximately 1400 patients with locally-advanced unresectable or metastatic gastric or gastroesophageal junction adenocarcinoma, who have received ramucirumab plus paclitaxel combination therapy will be collected.

DETAILED DESCRIPTION:
Ramucirumab plus paclitaxel combination therapy has shown a survival benefit in patients with previously treated gastric or gastroesophageal junction adenocarcinoma. However, the real-world efficacy and safety of ramucirumab plus paclitaxel combination therapy in Korea have only been evaluated once outside of controlled clinical trials. Therefore, this large multicenter retrospective analysis was designed to evaluate the real-world efficacy and safety of ramucirumab plus paclitaxel under the Korea National Health Insurance System. The medical records in approximately 1400 patients with locally-advanced unresectable or metastatic gastric or gastroesophageal junction adenocarcinoma, who have received ramucirumab plus paclitaxel combination therapy between May 2018 and December 2018 will be collected. Eligibility criteria included age ≥ 19 years, histologically or cytologically confirmed gastric or gastroesophageal junction adenocarcinoma, locally advanced unresectable or metastatic disease, and previous first-line systemic therapy including fluoropyrimidine and platinum. Efficacy was evaluated by overall survival, progression free survival, time to progression, objective response rate, disease control rate, and duration of response. Safety was evaluated by hematologic or non-non hematologic toxicities and adverse events of special interest with ramucirumab plus paclitaxel combination therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥19 years at the time of study registration
2. Histologically or cytologically confirmed gastric or gastroesophageal junction adenocarcinoma
3. Locally advanced unresectable or metastatic disease
4. Patients who have received previous palliative first-line systemic therapy including fluoropyrimidine and platinum for advanced gastric or gastroesophageal junction adenocarcinoma
5. Patients who have received ramucirumab plus paclitaxel combination therapy between May 2018 and December 2018 under the Korea National Health Insurance System

Exclusion Criteria:

1. Patients who have received ramucirumab plus paclitaxel combination therapy outside of the Korea National Health Insurance System
2. Patients who have received ramucirumab monotherapy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with locally-advanced unresectable or metastatic gastric or gastroesophageal junction adenocarcinoma, who have received ramucirumab plus paclitaxel combination therapy between May 2018 and December 2018 under the Korea National Health Insurance System
Sampling Method: Non-Probability Sample
Enrollment: 1063 (Actual)
Dates: Start 2019-12-18 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Overall survival | Until September 30, 2019
  Time from the start of ramucirumab plus paclitaxel to death from any cause
Progression free survival | Until September 30, 2019
  Time from the start of ramucirumab plus paclitaxel to disease progression or death from any cause
Incidence of adverse events | Until September 30, 2019
  Number (percentage) of subjects reporting adverse events

SECONDARY OUTCOMES:
Time to progression | Until September 30, 2019
  Time from the start of ramucirumab plus paclitaxel to disease progression
Objective response rate | Until September 30, 2019
  The proportion of subjects confirmed complete or partial response
Disease control rate | Until September 30, 2019
  The proportion of subjects confirmed complete or partial response or stable disease
Duration of response | Until September 30, 2019
  Time from documentation of tumor response to disease progression
Adverse events of special interest | Until September 30, 2019
  Number (percentage) of subjects reporting adverse events of special interest associated with ramucirumab plus paclitaxel

CONTACTS AND LOCATIONS:
Overall Officials: Dae Young Zang, Principal Investigator — Hallym University Medical Center
Locations (57):
- South Korea (57):
  - Korea University Ansan Hospital, Ansan
  - Hallym University Sacred Heart Hospital, Anyang
  - Soonchunhyang University Bucheon Hospital, Bucheon-si
  - The Catholic University of Korea, Bucheon ST. Mary's Hospital, Bucheon-si
  - Dongnam Institute of Radiological&Medical Sciences, Busan
  - Inje University Busan Paik Hospital, Busan
  - Dong-A University Hospital, Busan
  - Pusan National University Hospital, Busan
  - Kosin University Gospel Hospital, Busan
  - Samsung Changwon medical center, Changwon
  - Gyeongsang National University Changwon Hospital, Changwon
  - Dankook University Hospital, Cheonan
  - Soonchunhyang University Cheonan Hospital, Cheonan
  - Chungbuk National University Hospital, Cheonju
  - Kangwon National University Hospital, Chuncheon
  - Kyungpook National University Chilgok Hospital, Daegu
  - Yeungnam University Medical Center, Daegu
  - Keimyung University Dongsan Medical Center, Daegu
  - The Catholic University of Korea Daejeon ST. Mary's Hospital, Daejeon
  - Chungnam National University Hospital, Daejeon
  - Gangneung Asan Hospital, Gangneung
  - National Cancer Center, Goyang
  - Chosun University Hospital, Gwangju
  - Chonnam National University Hwasun Hospital, Hwasun
  - Wonkwang University Hospital, Iksan
  - The Catholic University of Korea Incheon ST. Mary's Hospital, Incheon
  - Gachon University Gil Medical Center, Incheon
  - Inha University Hospital, Incheon
  - Chonbuk National University Hospital, Jeonju
  - Gyeongsang National University Hospital, Jinju
  - Cha University Bundang Medical Center, Seongnam
  - Bundang Jesaeng Hospital, Seongnam
  - Seoul National University Bundang Hospital, Seongnam
  - Inje University Sanggye Paik Hospital, Seoul
  - Korea Cancer Hospital of Korea Institute of Radiological and Medical Sciences, Seoul
  - KyungHee University Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Soonchunhyang University Seoul Hospital, Seoul
  - Konkuk University Medical Center, Seoul
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Seoul ST. Mary's Hospital, Seoul
  - ChungAng University Hospital, Seoul
  - SMG-SNU Boramae Medical Center, Seoul
  - The Catholic University of Korea Yeouido ST. Mary's Hospital, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - The Catholic University of Korea ST. Mary's Hospital, Suwon
  - Ajou University Hospital, Suwon
  - The Catholic University of Korea Uijeongbu ST. Mary's Hospital, Uijeongbu-si
  - Ulsan University Hosiptal, Ulsan
  - Wonju Severance Christian Hospital, Wŏnju
  - Pusan National University Yangsan Hospital, Yangsan

REFERENCES:
- [Result] Jung KW, Won YJ, Kong HJ, Lee ES. Cancer Statistics in Korea: Incidence, Mortality, Survival, and Prevalence in 2016. Cancer Res Treat. 2019 Apr;51(2):417-430. doi: 10.4143/crt.2019.138. Epub 2019 Mar 18. PMID 30913865
- [Result] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Result] Wagner AD, Grothe W, Haerting J, Kleber G, Grothey A, Fleig WE. Chemotherapy in advanced gastric cancer: a systematic review and meta-analysis based on aggregate data. J Clin Oncol. 2006 Jun 20;24(18):2903-9. doi: 10.1200/JCO.2005.05.0245. PMID 16782930
- [Result] Bang YJ, Van Cutsem E, Feyereislova A, Chung HC, Shen L, Sawaki A, Lordick F, Ohtsu A, Omuro Y, Satoh T, Aprile G, Kulikov E, Hill J, Lehle M, Ruschoff J, Kang YK; ToGA Trial Investigators. Trastuzumab in combination with chemotherapy versus chemotherapy alone for treatment of HER2-positive advanced gastric or gastro-oesophageal junction cancer (ToGA): a phase 3, open-label, randomised controlled trial. Lancet. 2010 Aug 28;376(9742):687-97. doi: 10.1016/S0140-6736(10)61121-X. Epub 2010 Aug 19. PMID 20728210
- [Result] Kim HS, Kim HJ, Kim SY, Kim TY, Lee KW, Baek SK, Kim TY, Ryu MH, Nam BH, Zang DY. Second-line chemotherapy versus supportive cancer treatment in advanced gastric cancer: a meta-analysis. Ann Oncol. 2013 Nov;24(11):2850-4. doi: 10.1093/annonc/mdt351. Epub 2013 Aug 13. PMID 23942775
- [Result] Fuchs CS, Tomasek J, Yong CJ, Dumitru F, Passalacqua R, Goswami C, Safran H, Dos Santos LV, Aprile G, Ferry DR, Melichar B, Tehfe M, Topuzov E, Zalcberg JR, Chau I, Campbell W, Sivanandan C, Pikiel J, Koshiji M, Hsu Y, Liepa AM, Gao L, Schwartz JD, Tabernero J; REGARD Trial Investigators. Ramucirumab monotherapy for previously treated advanced gastric or gastro-oesophageal junction adenocarcinoma (REGARD): an international, randomised, multicentre, placebo-controlled, phase 3 trial. Lancet. 2014 Jan 4;383(9911):31-39. doi: 10.1016/S0140-6736(13)61719-5. Epub 2013 Oct 3. PMID 24094768
- [Result] Wilke H, Muro K, Van Cutsem E, Oh SC, Bodoky G, Shimada Y, Hironaka S, Sugimoto N, Lipatov O, Kim TY, Cunningham D, Rougier P, Komatsu Y, Ajani J, Emig M, Carlesi R, Ferry D, Chandrawansa K, Schwartz JD, Ohtsu A; RAINBOW Study Group. Ramucirumab plus paclitaxel versus placebo plus paclitaxel in patients with previously treated advanced gastric or gastro-oesophageal junction adenocarcinoma (RAINBOW): a double-blind, randomised phase 3 trial. Lancet Oncol. 2014 Oct;15(11):1224-35. doi: 10.1016/S1470-2045(14)70420-6. Epub 2014 Sep 17. PMID 25240821
- [Result] Smyth EC, Verheij M, Allum W, Cunningham D, Cervantes A, Arnold D; ESMO Guidelines Committee. Gastric cancer: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2016 Sep;27(suppl 5):v38-v49. doi: 10.1093/annonc/mdw350. No abstract available. PMID 27664260
- [Result] Muro K, Van Cutsem E, Narita Y, Pentheroudakis G, Baba E, Li J, Ryu MH, Zamaniah WIW, Yong WP, Yeh KH, Kato K, Lu Z, Cho BC, Nor IM, Ng M, Chen LT, Nakajima TE, Shitara K, Kawakami H, Tsushima T, Yoshino T, Lordick F, Martinelli E, Smyth EC, Arnold D, Minami H, Tabernero J, Douillard JY. Pan-Asian adapted ESMO Clinical Practice Guidelines for the management of patients with metastatic gastric cancer: a JSMO-ESMO initiative endorsed by CSCO, KSMO, MOS, SSO and TOS. Ann Oncol. 2019 Jan 1;30(1):19-33. doi: 10.1093/annonc/mdy502. PMID 30475956
- [Result] Japanese Gastric Cancer Association. Japanese gastric cancer treatment guidelines 2014 (ver. 4). Gastric Cancer. 2017 Jan;20(1):1-19. doi: 10.1007/s10120-016-0622-4. Epub 2016 Jun 24. No abstract available. PMID 27342689
- [Result] Guideline Committee of the Korean Gastric Cancer Association (KGCA), Development Working Group & Review Panel. Korean Practice Guideline for Gastric Cancer 2018: an Evidence-based, Multi-disciplinary Approach. J Gastric Cancer. 2019 Mar;19(1):1-48. doi: 10.5230/jgc.2019.19.e8. Epub 2019 Mar 19. No abstract available. PMID 30944757
- See also: NCCN Clinical Practive Guidelines in Oncology: Gastric Cancer. Version 1, 2019 — https://www.nccn.org/professionals/physician_gls/pdf/gastric.pdf